CLINICAL TRIAL: NCT06581224
Title: Implementation of a Primary Hospitalist Provider Team to Enhance the Care for High-Need High-Complexity Patients Requiring Hospitalization
Brief Title: Implementation of a Primary Hospital Provider (PHP) Team
Acronym: PHP Team
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-1299; A534270 (Other: UW Madison); Protocol Version 12/23/25 (Other: UW Madison)
Record Dates: First submitted 2024-08-29; First posted 2024-09-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: High-need, High-complexity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHP Team (Experimental): PHP Team
  Interventions: Other: Primary Hospital Provider Team
- Usual Care (No Intervention): Usual Care hospital medicine team

INTERVENTIONS:
Other: Primary Hospital Provider Team — The PHP team aims to enhance continuity during hospital readmissions with a consistent cohort of seven hospital medicine physicians and two advanced practice providers (APPs). To improve care transitions, the team will have an integrated case manager who will continue following PHP patients during subsequent hospitalizations. Physicians will follow a standard seven-day service schedule, with the two APPs alternating five-to-seven-day periods. Daily huddles between physicians and APPs will further promote continuity. During the index admission, the PHP team will create a care plan in consultation with the patient to improve standardization of inpatient care and transition to outpatient settings. Communication will be a core tenet of the team, with scheduled monthly team meetings of physicians, APPs, case manager, dyad partner, and representatives from nursing and therapy services to revise individualized care plans for PHP patients and brainstorm solutions for complex challenges.
  Arms: PHP Team

SUMMARY:
The goal of this pragmatic clinical trial is to learn if it is possible to implement a Primary Hospital Provider (PHP) team that aims to improve continuity of care for patients who are frequently hospitalized. The main question it aims to answer is: Are patients assigned to the PHP team more likely to be assigned to this team during a follow up hospitalization? Researchers will compare this to similar patients assigned to receive usual care. Some patient participants (or their caregivers) from both the PHP team and usual care groups will be asked to participate in interviews to help researchers understand the needs of patients who are frequently admitted and the care they receive.

DETAILED DESCRIPTION:
The overarching goal of this study is to reduce inpatient care fragmentation for high-need, high-complexity (HNHC) patients and improve outcomes by implementing a primary hospital provider (PHP) team. In this study, we will specifically evaluate the feasibility of implementation of this team as well as workforce and operational acceptance, as well as its impact on continuity of hospital medicine care across subsequent admissions.

The study is conducted as a two-arm, pragmatic hybrid type II effectiveness implementation trial with two sequential phases. Phase 1 focuses on initial feasibility and early acceptability of the PHP team. Phase 2 evaluates sustained implementation, reach, and longitudinal continuity outcomes using the same intervention, eligibility criteria, and study procedures. No changes will be made to the intervention, eligibility criteria, or data collection methods between phases.

Study Aims:

Aim 1 Primary Implementation Objective: Compare the fragmentation in hospital medicine care during subsequent admissions for HNHC patients assigned to the PHP team with those continuing to receive usual care.

* Aim 1a (Phase 1): Assess feasibility and early continuity of care during subsequent admissions.
* Aim 1b (Phase 2): Evaluate sustained continuity and re-exposure to the PHP team across repeated hospitalizations over an extended enrollment period.

Aim 2 Primary Exploratory Objective: Explore perceptions of care among HNHC patients and caregivers randomized to the PHP team and to a usual care team.

Aim 3 Secondary Exploratory Objective: Identify operational perceptions of the implementation of the PHP team from a workforce and system-level perspective.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 at the time of index admission
* Two or more hospitalizations to a general medicine service at UW Health (University Hospital or East Madison Hospital) within the past 12 months AND an EPIC Readmission Risk Score of greater than a predetermined value

Exclusion Criteria:

* Outpatient primary care provider is part of the UW Health Family Medicine service that currently admits their own patients to a separate service at University Hospital
* Patients with an oncologic diagnosis for which they are actively receiving chemotherapy or immunotherapy
* Incarcerated persons
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients readmitted to the PHP team | Implementation Phase 1 up to 9 months, Sustained Implementation Phase 2 up to 33 months
  The number of patients in the PHP arm who were readmitted to the PHP team on subsequent hospitalizations.
Number of patients readmitted to usual care team | Implementation Phase 1 up to 9 months, Sustained Implementation Phase 2 up to 33 months
  The number of patients in the usual care arm who were readmitted to a usual care team on subsequent hospitalizations.
Percentage of patients readmitted to the PHP team | Implementation Phase 1 up to 9 months, Sustained Implementation Phase 2 up to 33 months
  The percentage of patients in the PHP arm who were readmitted to the PHP team on subsequent hospitalizations.
Percentage of patients readmitted to usual care team | Implementation Phase 1 up to 9 months, Sustained Implementation Phase 2 up to 33 months
  The percentage of patients in the usual care arm who were readmitted to a usual care team on subsequent hospitalizations.

OTHER OUTCOMES:
Themes that emerge as barriers from the patient and/or caregiver perspective | 6 months
  Qualitative barriers during hospitalization for high-need, high-complexity patients that emerge from patient and/or caregiver interviews. Interviews will be coded and themed and reported here.
Themes that emerge as facilitators from the patient and/or caregiver perspective | 6 months
  Qualitative facilitators during hospitalization for high-need, high-complexity patients that emerge from patient and/or caregiver interviews. Interviews will be coded and themed and reported here.
Acceptability as assessed from the patient and/or caregiver perspective | 6 months
  Acceptability of the intervention will be assessed from patient and/or caregiver interviews. Interviews will be coded and themed and reported here
Themes that emerge as barriers from the hospitalist perspective | 4 months
  Qualitative barriers during hospitalization for high-need, high-complexity patients that emerge from focus groups with hospitalists. Focus groups will be coded and themed and reported here.
Themes that emerge as facilitators from the hospitalist perspective | 4 months
  Qualitative facilitators during hospitalization for high-need, high-complexity patients that emerge from focus groups with hospitalists. Focus groups will be coded and themed and reported here.
Acceptability as assessed from the hospitalist perspective | 6 months
  Acceptability of the intervention will be assessed from focus groups with hospitalists. Hospitalists will be coded and themed and reported here

CONTACTS AND LOCATIONS:
Overall Officials: Sara Westergaard, MD, MPH, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No